CLINICAL TRIAL: NCT00900094
Title: Proteomics Biomarker Development Laboratory (Aka IRB 1999-514)
Brief Title: UMCC 003 Cancer-Related Protein Biomarkers in Blood and Tumor Tissue of Patients With Cancer
Acronym: IRB 2000-294
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Dr. Dean Brenner, University of Michigan Comprehensive Cancer Center
Other Study IDs: CDR0000276589; U01CA084982 (NIH); P30CA046592 (NIH); CCUM-0003
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer; Colorectal Cancer; Esophageal Cancer; Liver Cancer; Lung Cancer; Ovarian Cancer; Pancreatic Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IV breast cancer; adenocarcinoma of the colon; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; adenocarcinoma of the pancreas; stage II pancreatic cancer; stage III pancreatic cancer; extensive stage small cell lung cancer; stage IIIC breast cancer; stage IV pancreatic cancer; recurrent breast cancer; recurrent colon cancer; recurrent esophageal cancer; recurrent non-small cell lung cancer; recurrent ovarian epithelial cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma; recurrent small cell lung cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Liver Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Carcinoma, Hepatocellular; Small Cell Lung Carcinoma | interventions — In Situ Hybridization, Fluorescence; Polymerase Chain Reaction; Immunohistochemistry; Mass Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: fluorescence in situ hybridization
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: mass spectrometry

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue in the laboratory from patients with cancer and blood from healthy participants may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at cancer-related protein biomarkers in the blood and tumor tissue of patients with cancer and in the blood of healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify tumor antigens that induce a humoral response in patients with cancer.
* Identify tumor-secreted proteins by special analysis in culture, and evaluate their expression patterns in tumors and preneoplastic lesions to further assess their potential specificity.
* Determine serum positivity and specificity of potential markers for early detection of cancer.

OUTLINE: This is a multicenter study.

Patients and healthy participants undergo blood collection. Patients with suspected or newly diagnosed disease undergo a second blood collection between 4-10 weeks after surgery (but before any additional cytotoxic therapy or radiotherapy) provided they had a surgical resection with negative margin. All patients are asked questions about family history of cancer, the development of their cancer, other medical history, past and present smoking history, and menstrual period for females.

DNA is extracted from the blood and from patient tumor tissue samples obtained during surgery. Immunohistochemistry (including polymerase chain reaction) and in situ hybridization are used to analyze protein expression patterns, after proteins are identified by mass spectrometry and amino acid sequencing.

PROJECTED ACCRUAL: A total of 3,150 patients and 1,200 healthy participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria (patient):

  * Scheduled to undergo primary surgical resection or first debulking surgery (prior to any anticancer treatment) for suspected or newly diagnosed cancer, including any of the following types:

    * Breast cancer
    * Adenocarcinoma of the colon
    * Adenocarcinoma or squamous cell carcinoma of the esophagus
    * Non-small cell lung cancer
    * Ovarian epithelial adenocarcinoma
  * Metastatic or unresectable cancer, including any of the following types:

    * Breast cancer
    * Adenocarcinoma of the colon
    * Adenocarcinoma or squamous cell carcinoma of the esophagus
    * Hepatoma
    * Non-small cell lung cancer
    * Small cell lung cancer
    * Ovarian epithelial adenocarcinoma
    * Adenocarcinoma of the pancreas
* Meets the following criteria (healthy participant):

  * No chronic disease

    * Healthy participants with a history of cancer must be cancer-free for 5 years (skin cancer or carcinoma in situ of the cervix within the past 5 years allowed)
  * Willing to provide 60 mL of blood
  * Not a blood relative of an eligible and consenting cancer patient

PATIENT CHARACTERISTICS:

* Able to tolerate the removal of 30-60 mL of blood
* No feelings of light-headedness, dizziness, or fainting within the past 2 weeks
* Pulse less than 100 on day of blood draw for study enrollment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy or radiotherapy for metastatic or unresectable cancer
* No concurrent chemotherapy
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The laboratory will apply technologies for protein analysis to the detection and identification of proteins secreted by tumor cells and protein antigens that induce a humoral response in tumors. The initial targeted tumor types for the identification of potential biomarker proteins are: Colon, esophagus, ovary, lung, breast and liver
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2000-06; Primary Completion 2006-12 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Identification of tumor antigens that induce a humoral response in cancer patients
Identification of tumor-secreted proteins by special analysis in culture
Tumor-secreted protein expression in tumors and preneoplastic lesions
Potential markers for early detection of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Samir M. Hanash, MD, PhD, Study Chair — University of Michigan Rogel Cancer Center